CLINICAL TRIAL: NCT01559285
Title: Effects of Epidurally Administered Ropivacaine Concentration on the Hemodynamic Parameters
Acronym: PNU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Assisstant Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PNU05-2011-054
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Epidural Anesthesia; Ropivacaine Concentration; Hemodynamics
Keywords: epidural, local, ropivacaine; epidural administration; stroke volume variability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.375% ropivacaine (Active Comparator): 0.375% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Interventions: Drug: 0.375% ropivacaine concentration
- 0.75% ropivacaine (Active Comparator): 0.75% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Interventions: Drug: 0.75% ropivacaine concentration
- 0.2% ropivacaine (Active Comparator): 0.2% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Interventions: Drug: 0.2% ropivacaine concentration

INTERVENTIONS:
Drug: 0.75% ropivacaine concentration — 0.75% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Arms: 0.75% ropivacaine
Drug: 0.375% ropivacaine concentration — 0.375% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Arms: 0.375% ropivacaine
Drug: 0.2% ropivacaine concentration — 0.2% ropivacaine 8ml was injected epidurally after induction of general anesthesia
  Arms: 0.2% ropivacaine

SUMMARY:
In this trial, the investigators intend to examine whether the concentration of local anesthetics during epidural analgesia could be modulating factor for change of hemodynamics in patients undergoing major upper abdominal surgery.

DETAILED DESCRIPTION:
One hundred and twenty patients scheduled for major abdominal surgery under TEA combined general anesthesia were randomized in a double-blinded method to receive one of three different concentration study solutions in 8 ml of volume after the induction of anesthesia: 0.75% ropivacaine (60 mg), 0.375% ropivacaine (30 mg), or 0.2% ropivacane (16 mg).

In each group, the patients were divided into two subgroups at the age of 60 to perform age based analysis. The acquired hemodynamic data after administration of epidural loading dose were compared and analyzed between young and elderly groups in each group.

ELIGIBILITY:
Inclusion Criteria: all of the followings needed.

* ASA I or II patients
* 18 to 65 years old
* undergoing major upper abdominal surgery
* planned combined thoracic epidural analgesia and general anesthesia

Exclusion Criteria:

* any contraindication to epidural analgesia
* allergy to local anesthetics of the amide type
* communication difficulties that would prevent reliable assessment
* known significant cardiac or respiratory disease
* pregnant
* patients who were not in cardiac sinus rhythm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2013-04-19 (Actual); Study Completion 2013-04-19 (Actual)

PRIMARY OUTCOMES:
hemodynamic changes depends on the concentration of ropivacaine | during 1hour after administration of epidural drug dosing
  Systolic blood pressure, diastolic blood pressure, MAP, HR, stroke volume, stroke volume, stroke volume index, stroke volume variation, cardiac output, and cardiac index were continuously measured at 5 minute intervals during 1 hour.

SECONDARY OUTCOMES:
Age based hemodynamic changes depends on the concentration of ropivacaine | during 1hour after administration of epidural drug dosing
  In each group, the patients were divided into two subgroups at the age of 60 to perform age based analysis. The acquired hemodynamic data after administration of epidural loading dose were compared and analyzed between young and elderly groups in each group.
  Systolic blood pressure, diastolic blood pressure, MAP, HR, stroke volume, stroke volume, stroke volume index, stroke volume variation, cardiac output, and cardiac index were continuously measured at 5 minute intervals during 1 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Jeong Lee, PhD, MD, Principal Investigator — Dept. of Anesthesia, Pusan National University, School of Medicine
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

REFERENCES:
- [Derived] Hong JM, Lee HJ, Oh YJ, Cho AR, Kim HJ, Lee DW, Do WS, Kwon JY, Kim H. Observations on significant hemodynamic changes caused by a high concentration of epidurally administered ropivacaine: correlation and prediction study of stroke volume variation and central venous pressure in thoracic epidural anesthesia. BMC Anesthesiol. 2017 Nov 16;17(1):153. doi: 10.1186/s12871-017-0444-x. PMID 29145824